CLINICAL TRIAL: NCT00208832
Title: A Randomized Controlled Trial to Improve Medication Compliance Among Patients With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 0784-2003; AHA 0335119N (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Disease
Keywords: Medication Compliance; Health Literacy
MeSH Terms: conditions — Coronary Disease; Medication Adherence

INTERVENTIONS:
Procedure: Graphic medication schedule (Pill card)
Procedure: Refill reminder postcard

SUMMARY:
Coronary heart disease (CHD) is the most common cause of death in the United States. A common term for CHD is "blocked arteries." People with CHD or "blocked arteries" often have high blood pressure, high cholesterol, or diabetes. They are also more likely to suffer a heart attack. Many heart attacks could be prevented by taking medicines that control blood pressure, cholesterol, and diabetes. However, only 50%-60% of patients take their medicines as directed. Patients who don't take their medicines regularly are considered noncompliant.

One of the risk factors for noncompliance is low health literacy. Health literacy is the ability to obtain, understand, and act on basic health information. Patients with low health literacy may not understand their illnesses as well, or how to take their medicines properly.

The purposes of this project are

1. to learn more about the relationship between low health literacy and medication compliance, and
2. to test 2 different strategies designed to help patients take their medicines more regularly.

Patients with CHD were recruited when they arrived for a regular doctor's appointment. We measured their health literacy skills, asked questions about how they take their medications, and checked their blood pressure and last cholesterol and diabetes measurements. We then assigned patients to 1 of 4 intervention groups (intervention ongoing). The first group is receiving usual care, which includes regular medication instructions printed on the bottle and no reminders to refill medicines. The second group gets monthly postcards reminding them to refill their prescriptions. The third group gets a new medication schedule that shows them, with pictures and figures, how they are supposed to take their medicines each day. The fourth group receives both the postcards and the new medication schedule. We are following patients for 1 year to see which intervention has the greatest impact on their medication compliance, blood pressure, cholesterol, and diabetes measurements. We will also examine whether patients' health literacy affects the success of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease, demonstrated by documentation of > 30% stenosis of one or more coronary vessels on cardiac catheterization, history of coronary artery bypass graft surgery, history of angioplasty, or documented myocardial infarction.

Exclusion Criteria:

* Current participation in another medication adherence study
* Too ill
* Does not manage their own medications
* No mailing address or telephone number
* Routine prescriptions filled outside of the Grady pharmacy system
* Psychiatric illnesses, overt delirium or dementia
* Visual acuity worse than 20/60
* Unable to communicate in English
* Already using a medication pill card

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2004-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Medication Compliance at one year

SECONDARY OUTCOMES:
Improved blood pressure, cholesterol, and diabetic control at one year

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Kripalani, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States